CLINICAL TRIAL: NCT01725009
Title: A Single-center, Open-label, Multiple-dose Study to Evaluate the Pharmacokinetics, Safety and Tolerability of Levetiracetam Administered as Intravenous Infusion in Japanese and Caucasian Healthy Male Subjects
Brief Title: Multiple-dose Study of Levetiracetam Injection in Japanese and Caucasian Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EP0038
Record Dates: First submitted 2012-11-07; First posted 2012-11-12 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Japanese; Caucasian
MeSH Terms: interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levetiracetam IV infusions in Japanese (Experimental): Multiple 15-minute intravenous infusions of 1500 mg levetiracetam in Japanese subjects
  Interventions: Drug: Multiple 15-minute intravenous infusions of 1500 mg levetiracetam
- Levetiracetam IV infusions in Caucasian (Experimental): Multiple 15-minute intravenous infusions of 1500 mg levetiracetam in Caucasian subjects
  Interventions: Drug: Multiple 15-minute intravenous infusions of 1500 mg levetiracetam

INTERVENTIONS:
Drug: Multiple 15-minute intravenous infusions of 1500 mg levetiracetam — Strength, 100 mg/mL; Form, concentrate for solution for infusion; Frequency, twice a day; Duration, 7 days
  Other Names: E-Keppra

SUMMARY:
To compare the pharmacokinetics of levetiracetam following single and multiple 15-minute intravenous infusions of 1500 mg levetiracetam between Japanese and Caucasian healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* healthy Japanese and Caucasian males with the age between 20 and 40 years old,
* with the body mass index between 20 and 25,
* with the body weight between 60 and 80kg

Exclusion Criteria:

* subjects who have a history or presence of drug addiction or excessive use of alcohol
* current smokers and former smokers who have given up since less than 6 months before the first dose
* heavy caffeine drinker

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration after a single dose (Cmax) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of Intravenous (IV) infusion
Area under the curve from zero to the time of the last quantifiable concentration after a single (AUC(0-t)) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion
Area under the plasma concentration time curve from zero to infinity after a single dose (AUC) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion
Body-weight normalized maximum plasma concentration after a single dose (Cmax) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion
Body-weight normalized area under the curve from zero to the time of the last quantifiable concentration after a single, (AUC(0-t)) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion
Body weight normalized area under the plasma concentration time curve from zero to infinity after a single dose, (AUC) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion
Maximum plasma concentration at steady state after multiple doses (Cmax,ss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.
Area under the curve over a dosing interval at steady state after multiple doses (AUCτss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.
Body-weight normalized maximum plasma concentration at steady state after multiple doses (Cmax,ss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.
Body-weight normalized area under the curve over a dosing interval at steady state after multiple doses (AUCτss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.

SECONDARY OUTCOMES:
Area under the curve over a dosing interval, (AUCτ (τ = 12 hours)) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion
Time to maximum plasma concentration after a single dose (tmax) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
Terminal elimination half-life after a single dose (t1/2) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
First order terminal elimination rate constant after a single dose (λz) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
Total body clearance after a single dose (CL) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
Volume of distribution during terminal phase after a single dose (Vz) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
Mean residence time after a single dose (MRT) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of IV infusion.
Time to maximum plasma concentration at steady state after multiple doses (tmax,ss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.
Total body clearance at steady state after multiple doses (CLss) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of IV infusion.
Linearity factor after multiple doses (LF) | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9, 12, 24 and 36 hours after the start of the first IV infusion and at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of the last IV infusion.
  LF = AUCτss / AUC
Accumulation ratio (RAUC) after multiple doses | Multiple samples at predose, 5, 10, 15, 30, 45 minutes, 1, 1.5, 2, 3, 6, 9 and 12 hours after the start of the first and the last IV infusions
  RAUC = AUCτss / AUCτ

CONTACTS AND LOCATIONS:
Locations (1):
- 01, Tokyo, Japan